CLINICAL TRIAL: NCT00547482
Title: The TANTALUS® II System for the Treatment of Type 2 Diabetes: A Randomized Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol design under review.
Sponsor: MetaCure (USA), Inc. (Industry)
Responsible Party: MetaCure (USA) Inc., MetaCure (USA), Iinc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MC CR TAN2006-067
Record Dates: First submitted 2007-10-04; First posted 2007-10-22 (Estimated); Last update posted 2010-12-16 (Estimated); Status verified 2008-04

CONDITIONS: Type 2 Diabetes Mellitus; Overweight
Keywords: Type 2 Diabetes; Overweight; Obese
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity | interventions — Drug Delivery Systems

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Sham Comparator): They will all be implanted but not activated for the Initial Study Period (24 weeks), followed by all subjects assigned to treatment (Control Group with device activation) in the Study Extension Period (an additional 24 weeks). Subjects will remain in the study (Safety Monitoring Period) with semi-annual evaluations until a determination of safety and efficacy is made by the FDA.
  Interventions: Device: TANTALUS(TM) System
- Treatment (Active Comparator): All subjects will be implanted with the TANTALUS System (IPG with Charge Coil and UltraFlex leads) and randomized into either the "Treatment Group" or "Control Group" after surgery at Week 1, Visit 5 (device activation). They will be followed for the Initial Study Period (24 weeks), followed by the Study Extension Period (an additional 24 weeks). Subjects will remain in the study (Safety Monitoring Period) with semi-annual evaluations until a determination of safety and efficacy is made by the FDA.
  Interventions: Device: TANTALUS(TM) System

INTERVENTIONS:
Device: TANTALUS(TM) System — All subjects will be implanted with the TANTALUS System (IPG with Charge Coil and UltraFlex leads) and randomized into either the "Treatment Group" or "Control Group" after surgery at Week 1, Visit 5 (device activation).

SUMMARY:
The main purpose of this research study is to investigate whether the TANTALUS II System is effective in improving glycemic (blood sugar) control in subjects who have type 2 diabetes (high blood sugar) and are overweight. The research will also evaluate the impact on weight loss and will study other health conditions related to obesity.

This research study involves an experimental system. The experimental system is the TANTALUS System, which consists of the implantable portion that includes the implantable pulse generator (IPG) and three pairs of implantable leads. There are also three external parts (items that are used outside your body): the programmer, the charger, and the Patient Wand.

DETAILED DESCRIPTION:
This is a randomized, double-blind and controlled, multi-center study. Three hundred (300) subjects with type 2 diabetes ranging from low BMI to BMI 45 (BMI ≥ 28 and ≤ 45) will be enrolled.

The duration of subject participation in the main portion of the study which includes the initial study and study extension periods is expected to be approximately 12 months. Upon completion of this period, subjects with a TANTALUS device shall continue to be followed clinically at six-month intervals (Safety Monitoring Period) until the FDA has made a determination regarding the safety and efficacy of the device.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) ≥ 28 and ≤ 45 (kg/m2)
2. Type 2 diabetes >6 months
3. Type 2 diabetic subjects treated with oral anti-diabetic
4. Stable anti-diabetic medications ≥3 months prior to enrollment, six months for TZD
5. HbA1c ≥7.5% and ≤ 9.5 % at Visit 1, subjects with T2DM duration > 10 yrs should have HbA1c ≥7.5% and ≤ 9.0
6. Stable HbA1c, Stable weight, and stable treatment with anti-hypertensive and/or lipids lowering medications
7. Fasting blood glucose >120 and < 240 mg/dl at Visit 1, subjects with T2DM duration > 10 yrs should be >120 and ≤180.
8. Women with childbearing potential must agree to use adequate birth control methods
9. Stable weight - no significant change (variation < 5%) in the last 6 months
10. Willingness to perform at least 4 capillary blood glucose tests per day twice a week for the duration of the study
11. Willingness to refrain from using prescription, over the counter or herbal weight loss products for the duration of the trial
12. Ability and willingness to perform required study and data collection procedures and adhere to operating requirements of the TANTALUS II System
13. Alert, mentally competent,
14. Able to provide voluntary informed consent and HIPAA Authorization

Exclusion Criteria:

1. Receiving insulin therapy
2. Taking GLP-1, Amylin treatment (Byetta, Symlin)
3. Blood pressure levels of >180/100
4. Patients with an EF less than 35% (obtained within last 6 months) or indicated for an ICD; if echocardiogram outdated or unavailable, procedure to be done
5. Taking medications known to affect gastric motility such as narcotics (chronic use) and anticholinergics/antispasmodics
6. Use of prescription, over the counter or herbal weight loss products or obesity drugs during the two months prior to enrollment
7. Experiencing severe and progressing diabetic complications (i.e. retinopathy not stabilized, nephropathy with macroalbuminuria)
8. Prior wound healing problems due to Staphylococcus and Candida
9. Prior bariatric surgery
10. History of pancreatitis
11. History of peptic ulcer disease within 5 years of enrollment
12. Diagnosed with gastroparesis
13. Use of active medical devices (either implantable or external) such as ICD, pacemaker, neurostimulator (either implanted or worn). Subjects using an external active device who are able and willing to avoid use of the device during the study may be enrolled.
14. Cardiac history that physician feels should exclude the patient
15. Use of another investigational device or agent in the 30 days prior to enrollment
16. A history of life-threatening disease within 5 years of enrollment
17. Any additional condition(s) that in the Investigator's opinion would warrant exclusion from the study or prevent the subject from completing the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2007-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Glycemic control as measured by HbA1c: Difference in mean reduction between Control and Treatment Groups will be evaluated. | At the end of the Initial Study Period

SECONDARY OUTCOMES:
Device/procedure-related adverse events;hypoglycemic events; Proportion of subjects with HbA1c less than 7.0;reduction of weight for both groups;improvement of glycemic control as measured by HbA1c | The end of the Initial Study Period

CONTACTS AND LOCATIONS:
Overall Officials: Harold Lebowitz, MD, Study Chair — Professor of Medicine, Endocrinology and Metabolism/Diabetes, State University of NY Health Science
Locations (10):
- United States (10):
  - Scripps Clinic Del Mar, La Jolla / San Diego, California
  - Cedars Sinai, Los Angeles, California
  - University of Colorado at Denver Health Sciences Center, Denver, Colorado
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Kaleida Health, Diabetes-Endocrinology Center of Western New York, Buffalo, New York
  - Comprehensive Weight Control Program Cornell Medical Center, New York, New York
  - Mt. Sinai School of Medicine, New York, New York
  - University of Pennsylvania, Pennsylvania, Pennsylvania
  - Vanderbilt University School of Medicine, Nashville, Tennessee
  - Diabetes and Glandular Disease Clinic (DGD), San Antonio, Texas

REFERENCES:
- [Background] Peles S, Petersen J, Aviv R, Policker S, Abu-Hatoum O, Ben-Haim SA, Gutterman DD, Sengupta JN. Enhancement of antral contractions and vagal afferent signaling with synchronized electrical stimulation. Am J Physiol Gastrointest Liver Physiol. 2003 Sep;285(3):G577-85. doi: 10.1152/ajpgi.00109.2003. Epub 2003 Jun 11. PMID 12801883
- [Result] Bohdjalian A, Prager G, Aviv R, Policker S, Schindler K, Kretschmer S, Riener R, Zacherl J, Ludvik B. One-year experience with Tantalus: a new surgical approach to treat morbid obesity. Obes Surg. 2006 May;16(5):627-34. doi: 10.1381/096089206776945101. PMID 16687033
- See also: Related Info — http://www.metacure.com